CLINICAL TRIAL: NCT03795506
Title: Temperature Controlled Laminar Airflow (TLA) Treatment of Moderate to Severe Atopic Eczema in Children and Adolescents - a Randomized Placebo Controlled Phase 2 Study
Brief Title: TLA in Children With Moderate to Severe Atopic Eczema (TLA4AE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: JP Moulton Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18SM4747
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Atopic Dermatitis Eczema
Keywords: Atopic Dermatitis Eczema
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TLA Device (Experimental): 12 week overnight treatment with the active Temperature Controlled Laminar Airflow device.
  Interventions: Device: Nocturnal Temperature controlled Laminar Airflow (TLA) Treatment
- Placebo TLA Device (Placebo Comparator): 12 week overnight treatment with the placebo Temperature Controlled Laminar Airflow device.
  Interventions: Device: Placebo TLA Device

INTERVENTIONS:
Device: Nocturnal Temperature controlled Laminar Airflow (TLA) Treatment — 12 weeks of overnight treatment with active TLA device
  Arms: Active TLA Device
Device: Placebo TLA Device — 12 weeks of overnight use of placebo TLA device
  Arms: Placebo TLA Device

SUMMARY:
This is a single centre randomised, placebo-controlled phase 2 study in which 96 children age 4 to 16 years with moderate to severe, longstanding allergic eczema will be enrolled.

DETAILED DESCRIPTION:
Following a 4 to 6 week period on standardised treatment (run-in period, to ensure everyone starts with the same treatment approach), participants will be randomised to an active or dummy temperature-controlled laminar airflow (TLA) device, which has been shown to markedly reduce exposure to particles which can cause allergic reactions when being inhaled (inhaled allergens) and other particles which are in the air the investigators breathe in. This has been shown to be an effective treatment of atopic asthma.

The participants will undergo a 12-week treatment period. The device will then be removed and a final follow-up visit occurs at 16 weeks. The total study duration, including the run-in period is up to 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 16 years at time of consent
* Persistent moderate to severe eczema despite treatment with topical corticosteroids (TCS) Class II or more and/or topical calcineurin inhibitors (TCI, licenced use only) for at least 3 months.
* Eczema Area and Severity Index (EASI) Score ≥12 at screening and randomisation visit and >10% body surface involved
* Sensitisation to house dust mite species, confirmed by specific Immunoglobulin E (ImmunoCAP ≥2) and/or Skin Prick Test (SPT ≥5mm)
* Child able to sleep in their own bed and able to use the device for at least 5 out of 7 nights per week
* Written, informed consent of parent/legal guardian and patient assent

Exclusion Criteria:

* very severe atopic dermatitis
* use of systemic immunosuppression (such as cyclosporine, methotrexate, azathioprine, oral steroids) or UV therapy or extracorporal photopheresis within four weeks prior to the screening visit
* received therapeutic monoclonal antibodies (such as Omalizumab or Dupilumab) within six months prior to the screening visit
* Ongoing or planned desensitisation / immunotherapy during the study
* Infections requiring systemic antimicrobial treatment within four weeks prior to the screening visit
* Introduction of special dietary restriction (for eczema treatment) within three months prior to screening visit
* Severe asthma ≥ Step 4 and/or ≥1 course of systemic oral steroids for asthma in the three months prior to screening visit
* Significant underlying chronic medical condition (chronic other skin disease, inflammatory bowel disease, immunodeficiencies, other uncontrolled systemic disease, cancer)
* Planned time away from home (=unable to use TLA) exceeding 2 days/week; unable to use the device at least 5/7 days in the 2-3 weeks prior to end of intervention period.
* Prior research participation is not an exclusion criterion, except if it involved eczema disease modifying agents.
* Participating in current research

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of eczema severity (Eczema Area Severity Index = EASI Score, total) at week 12 compared to baseline | 12 weeks
  Change of eczema severity (EASI Score) at week 12 compared to baseline; higher score = higher severity. range 0-72 (0=no eczema, 72 highest severity)

SECONDARY OUTCOMES:
(Eczema Area Severity Index = EASI): EASI 50, EASI 75 | 12 weeks
  Proportion of participants achieving at least a 50% (EASI 50) or 75% (EASI 75) reduction of eczema severity. EASI range 0-72 (0=no eczema, 72 highest severity)
Change in SCORing Atopic Dermatitis = SCORAD Index | 12 weeks
  Change in total SCORAD Index at week 12 compared to baseline; higher score = higher severity; range 0-103 (0=no eczema, 103 highest severity)
Proportion of subjects achieving Investigator Global Assessment (IGA) of 0 or 1 | 12 weeks
  Proportion of subjects achieving Investigator Global Assessment (IGA) of 0 or 1; maximum score is 5 = most severe
Change in health related quality of life [QoL] from baseline for participants: CDQLI | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change in health related quality of life during run-in period, 12 week treatment period and 4 weeks after treatment end using Children's Dermatitis Quality of Life Index (CDQLI). Range 0-30 (0=no QoL impairment, 30 severe QoL impairment)
Improvement of itch; Visual Analogue Score (VAS), from baseline | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change of itch intensity during during run-in period, 12 week treatment period; and 4 weeks after treatment end; Visual Analogue Score (VAS) range 0-100; higher score = higher severity
Improvement of sleep; Visual Analogue Score (VAS), from baseline | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change of sleep disturbance during run-in period, 12 week treatment period and 4 weeks after treatment end; Visual Analogue Score (VAS) range 0-100; higher score = higher severity
Change in adverse impact on participants' families from baseline | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change in adverse impact of participants' eczema on families,during run-in period, 12 week treatment period and 4 weeks after treatment end using Dermatitis Family Impact Questionnaire (DFI); higher score = worse impact. Range 0-30 (0=no impact, 30 severe adverse impact)
Change of patient reported eczema activity from baseline | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change of patient reported eczema activity during run-in period, 12 week treatment period and 4 weeks after treatment end, using Patient Oriented Eczema Measure (POEM) tool; total score reported, higher score = higher severity; Range 0-28 (0=no impairment, 28 severe reported eczema symptoms)
Change in medication requirements (topical immunomodulators) from baseline | 20-22 weeks (baseline 4-6 weeks, intervention 12 weeks, 4 weeks after intervention)
  Change in medication requirements during run-in period, 12 week treatment period and 4 weeks after treatment end (topical immunomodulators, topical steroids, topical calcineurin inhibitors) from baseline
Change in sleep quality from baseline: actigraphy | 4-6 weeks
  Change in sleep quality, measured by actigraphy before and in first month after intervention start (total movement activity reported, higher scores = worse sleep disturbance); this is not a limited scale but simply counts the number of times an individual moves.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gore, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- IMPERIAL COLLEGE HEALTHCARE NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gore C, Gore RB, Fontanella S, Haider S, Custovic A. Temperature-controlled laminar airflow (TLA) device in the treatment of children with severe atopic eczema: Open-label, proof-of-concept study. Clin Exp Allergy. 2018 May;48(5):594-603. doi: 10.1111/cea.13105. Epub 2018 Mar 13. PMID 29383776
- [Background] Gore RB, Boyle RJ, Gore C, Custovic A, Hanna H, Svensson P, Warner JO. Effect of a novel temperature-controlled laminar airflow device on personal breathing zone aeroallergen exposure. Indoor Air. 2015 Feb;25(1):36-44. doi: 10.1111/ina.12122. Epub 2014 Jun 10. PMID 24750266
- [Background] Spilak MP, Sigsgaard T, Takai H, Zhang G. A Comparison between Temperature-Controlled Laminar Airflow Device and a Room Air-Cleaner in Reducing Exposure to Particles While Asleep. PLoS One. 2016 Nov 29;11(11):e0166882. doi: 10.1371/journal.pone.0166882. eCollection 2016. PMID 27898693
- [Background] Boyle RJ, Pedroletti C, Wickman M, Bjermer L, Valovirta E, Dahl R, Von Berg A, Zetterstrom O, Warner JO; 4A Study Group. Nocturnal temperature controlled laminar airflow for treating atopic asthma: a randomised controlled trial. Thorax. 2012 Mar;67(3):215-21. doi: 10.1136/thoraxjnl-2011-200665. Epub 2011 Nov 30. PMID 22131290